CLINICAL TRIAL: NCT03626272
Title: Effects of the Periodic Application of in Situ Simulation in Cardiopulmonary Resuscitation: Randomized Controlled Trial.
Brief Title: Effects of the in Situ Simulation to Competencies in Cardiopulmonary Resuscitation in the Nursing Team.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federal University of Health Science of Porto Alegre (Other)
Responsible Party: Principal Investigator, Cleidilene Ramos Magalhães, Principal Investigator, Federal University of Health Science of Porto Alegre
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: UFCSPA33
Record Dates: First submitted 2018-03-08; First posted 2018-08-13 (Actual); Last update posted 2018-08-13 (Actual); Status verified 2018-08

CONDITIONS: Learning Disorders
MeSH Terms: conditions — Learning Disabilities | interventions — Early Intervention, Educational

STUDY DESIGN:
Intervention Model Description: This is a randomized, non-blind controlled trial that will compare three periodicities of an educational intervention to be performed through in situ simulation. Group A will be submitted to intervention at 8-month intervals, group B every four months and group C every two months; each group will be divided into two subgroups, totaling six subgroups consisting of one nurse and three nursing technicians.
  The research was approved by the Research Ethics Committees of the Federal University of Health Sciences of Porto Alegre, under approval certificate no. 56516216.9.0000.5345, and of the Universidade Católica do Rio Grande do Sul/PUCRS, under approval certificate no. 56516216.9.3001.5336.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 8-month intervals (Active Comparator): Participants will be submitted to the educational intervention with in situ simulation every 8 months.
  Interventions: Other: educational intervention
- 4-month intervals (Active Comparator): Participants will be submitted to the educational intervention with in situ simulation every 4 months.
  Interventions: Other: educational intervention
- 2-month intervals (Active Comparator): Participants will be submitted to the educational intervention with in situ simulation every 2 months.
  Interventions: Other: educational intervention

INTERVENTIONS:
Other: educational intervention — The simulation scenarios were constructed using the service environment, with real equipment and materials and a low fidelity mannequin. The interventions were not filmed, and the clinical cases elaborated were fictitious, with clear objectives and developed according to the context of the unit. The simulations took place during the working hours of the participants, with the expected duration of the 10 minutes (average) for the scenario, and the average duration of the debriefing was 10 minutes, which took place immediately after the simulation and in the same location of the scenario.

SUMMARY:
Introduction: In situ simulation is a methodology that meets the concept of permanent education, since it allows learning from the context of practice and in the work environment itself.

Objective: to compare the development of skills (knowledge and skills) for CPR between groups submitted to different in situ simulation periodicities, and to identify the level of confidence to participate in a CPR.

Method: A randomized controlled, non-blind study comparing 3 periodicities of educational intervention performed by in situ simulation. This study will include nursing professionals from the nephrology department of a university hospital. The sample will be composed of 24 randomized participants in the groups, using opaque envelopes for each periodicity of training and professional category, being subdivided into 3 groups of periodicities with intervals of 2, 4 and 8 months. The instruments will evaluate the knowledge and skills in cardiopulmonary resuscitation and the perception of preparation for performing the maneuvers.

DETAILED DESCRIPTION:
The objective is to compare the development of skills (knowledge and skills) for CPR between groups submitted to different in situ simulation periodicities, and to identify the level of confidence to attend a CPR.

ELIGIBILITY:
Inclusion Criteria:

* They must be nurses and nursing technicians.

Exclusion Criteria:

* not complete the evaluations
* be under 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-11 (Estimated); Study Completion 2019-08 (Estimated)

PRIMARY OUTCOMES:
Average number of hits in the test of knowledge on cardiopulmonary resuscitation | up to eight months
  Measurement of the average/median/standard deviation of hits in the questions of the knowledge test, in each group (A, B, C,). This measurement was performed in two moments:
  * Pre and post initial intervention: measure performed to evaluate the impact of the initial intervention on the participants' knowledge about the issue.
  * After simulation intervention: measurement performed to evaluate the impact of the simulation intervention on the maintenance of knowledge, according to the periodicity group of intervention where the participant was allocated.
  The measurement was applied to all groups at the same moments. The following tests were used to make comparisons among groups: Wilcoxon Test; Estimate of the size of the Cohen's d effect (paired data); Kruskal-Wallis Test - Dunn's Post Hoc; Cohen's d: Effect size measures by the " Cohen's d" method complemented by the Confidence Interval 95%.
Average number of hits in the accomplishment of a set of skills. | Group A was evaluated when receiving the intervention every eight months, group B every four months, and group C every two months.
  To compare, among groups exposed to the periodicity of different interventions, the average/median/standard deviation of hits in the accomplishment of a set of skills that matches the CPR procedures. Group A was evaluated when receiving the intervention every eight months, group B every four months, and group C every two months.
  The Kruskal-Wallis Test was applied to compare the significance of the average outcomes among groups.
Average agreement in the preparation for CPR | up to eight months
  To Measure the average/median/standard deviation, referring to the agreement level of preparation for the accomplishment of CPR, in order to check the impact of the intervention performed according to the periodicity of application.
  The following tests were used to make comparisons among groups: Wilcoxon Test; Estimate of the size of the Cohen's d effect (paired data); Kruskal-Wallis Test - Dunn's Post Hoc; Cohen's d: Effect size measures by the "Cohen's d" method complemented by the Confidence Interval 95%.

CONTACTS AND LOCATIONS:
Locations (1):
- Cleidilene Ramos Magalhaes, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: Undecided